CLINICAL TRIAL: NCT06811844
Title: Comparison of Two-cycle and Three-cycle Induction Therapy With Modified TPF Regimen Combined and Camrelizumab for Locally Advanced Nasopharyngeal Carcinoma: A Prospective, Phase II, Multicenter, Randomized Controlled Study
Brief Title: Two-cycle and Three-cycle Induction Therapy With Modified TPF Regimen Combined and Camrelizumab for LANPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, San-Gang Wu, Clinical professor, The First Affiliated Hospital of Xiamen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XMYY-2024KY230-03
Record Dates: First submitted 2025-01-25; First posted 2025-02-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Nasopharyngeal Neoplasms; PD-1 Inhibitor; Induction Therapy; Complete Response; Chemotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Pathologic Complete Response | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two-cycle (Experimental): Two cycles induction chemotherapy + immunotherapy
  Interventions: Drug: Two-cycle induction chemotherapy + immunotherapy
- Three-cycle (Active Comparator): Three cycles induction chemotherapy + immunotherapy
  Interventions: Drug: Three-cycle induction chemotherapy + immunotherapy

INTERVENTIONS:
Drug: Two-cycle induction chemotherapy + immunotherapy — Two cycles of nab-paclitaxel at 260 mg/m2 on day 1, cisplatin at 25 mg/m2 from days 1 to 3, and oral S1 twice daily from days 1 to 14 (40 mg twice daily on patients with a body surface area [BSA] less than 1.25 m2, 50 mg twice daily for patients with a BSA between 1.25 and 1.5 m2, and 60 mg twice daily for patients with a BSA >1.5 m2). Camrelizumab was administered intravenously at a dose of 200 mg on the first day of each cycle.
  Other Names: 2
  Arms: Two-cycle
Drug: Three-cycle induction chemotherapy + immunotherapy — Three cycles of nab-paclitaxel at 260 mg/m2 on day 1, cisplatin at 25 mg/m2 from days 1 to 3, and oral S1 twice daily from days 1 to 14 (40 mg twice daily on patients with a body surface area [BSA] less than 1.25 m2, 50 mg twice daily for patients with a BSA between 1.25 and 1.5 m2, and 60 mg twice daily for patients with a BSA >1.5 m2). Camrelizumab was administered intravenously at a dose of 200 mg on the first day of each cycle.
  Other Names: 3
  Arms: Three-cycle

SUMMARY:
This prospective, phase II, multicenter, randomized controlled study aims to compare the complete response rate and long-term survival outcomes of two-cycle and three-cycle induction therapy with modified TPF regimens combined with camrelizumab in patients with locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Currently, the recommended number of cycles for induction chemotherapy in nasopharyngeal carcinoma primarily suggests two-three cycles of induction therapy. However, several studies have found that three cycles of induction therapy did not improve patient survival and may further increase hematological toxicity and gastrointestinal toxicity compared to those treated with two cycles of induction therapy. Based on research from our center, three cycles of induction therapy also did not improve patient survival. The latest 2024 CSCO guidelines have recommended that immunotherapy can be incorporated into the induction therapy stage for locally advanced nasopharyngeal carcinoma. Therefore, based on these research findings, the investigators hypothesize that two cycles of induction chemotherapy combined with immunotherapy will not be inferior to three cycles in terms of tumor response rates and may have lower adverse reactions. The investigators aim to compare the complete response rates and long-term survival outcomes of two-cycle and three-cycle modified TPF regimens combined with camrelizumab in patients with locally advanced (T1-4N2-3M0) nasopharyngeal carcinoma, providing new options for toxicity-reduced treatment in nasopharyngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old;
* Pathologically (including histology or cytology) confirmed nasopharyngeal carcinoma patients, with clinical staging T1-4N2-3M0 (according to the UICC/AJCC TNM staging system, 8th edition);
* No prior systemic treatment (surgery, radiotherapy, chemotherapy, etc.);
* At least one measurable lesion on imaging (as per RECIST criteria version 1.1);
* ECOG Performance Status (PS): 0-1;
* Expected survival ≥3 months;
* Male subjects and women of childbearing potential must use contraception from the first dose of study medication until 24 weeks after the last dose of study medication;
* Normal major organ function, with basic normal results in hematology, biochemistry, and coagulation tests;
* The investigator believes that the treatment will provide a survival benefit.

Exclusion Criteria:

* Active, known, or suspected autoimmune disease;
* Patients with hypertension that cannot be controlled to normal range despite antihypertensive medication (systolic BP >160 mmHg, diastolic BP >90 mmHg);
* History of hereditary bleeding tendency or coagulation dysfunction. Any clinically significant bleeding symptoms within 12 weeks prior to screening, or cumulative bleeding over 50 ml in 24 hours;
* Unwell-controlled cardiac clinical symptoms or diseases;
* Interstitial lung disease, drug-induced pneumonia, steroid-treated radiation pneumonitis, active pneumonia with symptoms, or severe pulmonary dysfunction;
* Active hepatitis B (HBV DNA ≥2000 IU/mL or 10^4 copies/mL), hepatitis C (HCV antibody positive and HCV-RNA above the lower limit of detection of the assay);
* Allergy to any of the study drugs;
* Pregnant or breastfeeding women;
* Any other factors that, in the investigator's judgment, may cause premature termination of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response | At the end of Cycle 2 or Cycle 3 (each cycle is 21 days)
  Complete Remission after induction therapy means that all detectable signs of the tumor have disappeared, including all measurable and assessable diseases. This includes the absence of any tumor lesions in imaging studies.

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival was measured from the day of the NPC diagnosis until disease recurrence and death from any cause.
Overall survival | 3 years
  Overall survival was measured from the day of the NPC diagnosis until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhangzhou Affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian
  - Hainan General Hospital, Haikou, Hainan

IPD SHARING:
Plan to Share IPD: No